CLINICAL TRIAL: NCT03932123
Title: Efficacy and Safety of Antibiotics in the Treatment of Early Onset Neonatal Sepsis
Brief Title: Antibiotic Therapy for Early Onset Neonatal Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: Tianjin Central Hospital of Gynecology Obstetrics (Other); Shandong Provincial Hospital (Other Government); Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhao, Head of department of clinical pharmacy and pharmacology, Shandong University
Other Study IDs: 2019_EOS_001
Record Dates: First submitted 2019-04-24; First posted 2019-04-30 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Early Onset Neonatal Sepsis
MeSH Terms: conditions — Neonatal Sepsis | interventions — Piperacillin; Tazobactam; Azlocillin; Moxalactam; Meropenem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Piperacillin and tazobactam, azlocillin, latamoxef, meropenem, vancomycin，cefotaxime — Efficacy and safety of antibiotics

SUMMARY:
Antibiotic therapy for early onset neonatal sepsis recommended by international guidelines and relevant studies is only kind of treatment regimen that penicillin G/ penicillin/ampicillin combined with gentamicin as the first-line treatment regimen. However, it is not applicable to the clinical practice in many countries and regions. We aim to study efficacy and safety of antibiotics in the treatment of early onset neonatal sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Age: postnatal age ≤ 72h;
* Meets NICE guidelines for using antibiotics to treat EONS;
* Azlocillin used as part of antimicrobial treatment;
* Parental written consent.

Exclusion Criteria:

* Expected survival time less than the treatment cycle;
* Major congenital malformations;
* Undergoing surgery within the first week of life;
* Receiving other systemic trial drug therapy;
* Other factors that the researcher considers unsuitable for inclusion.

Ages: 0 Days to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates suffered from early onset neonatal sepsis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-05-05 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | 72 hours after ending initial antibiotic therapy
  * requiring additional courses of antibiotic therapy within 72 hours after ending initial antibiotic therapy and/or
  * progression of the illness, necessitating a change of antibiotic and/or
  * blood culture isolate reported resistant to the antibiotic.

SECONDARY OUTCOMES:
Treatment duration | Through study completion, an average of 3 days
  Duration of initial antibiotic therapy
Duration of hospitalization | In the first month of patients' life
  Duration of hospitalization of patients
PD target | Through study completion, an average of 3 days
  The time of free drug concentration exceeding the minimal inhibitory concentration (fT>MIC)
White blood cell count | Through study completion, an average of 3 days
  White blood cell count in ×10^9/L
Procalcitonin | Through study completion, an average of 3 days
  Procalcitonin in ng/mL
C-reactive protein | Through study completion, an average of 3 days
  C-reactive protein in mg/L
Death | In the first month of patients' life
  Death in the first month of life
Adverse events | Through study completion, an average of 3 days
  Drug-related adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Central Hospital of Gynecology Obstetrics, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Wu YE, Wang T, Yang HL, Tang BH, Kong L, Li X, Gao Q, Li X, Yao BF, Shi HY, Huang X, Wang WQ, Jacqz-Aigrain E, Allegaert K, van den Anker J, Tian XY, Zhao W. Population pharmacokinetics and dosing optimization of azlocillin in neonates with early-onset sepsis: a real-world study. J Antimicrob Chemother. 2021 Feb 11;76(3):699-709. doi: 10.1093/jac/dkaa468. PMID 33188385